CLINICAL TRIAL: NCT07371728
Title: Effect of Aprepitant on Post-operative Nausea and Vomiting in Otologic Surgery: A Pilot Randomized-Controlled Trial
Brief Title: Effect of Aprepitant on Post-operative Nausea and Vomiting in Otologic Surgery
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Emily Kay-Rivest, Otolaryngologist, Sir Mortimer B. Davis - Jewish General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2026-4646
Record Dates: First submitted 2026-01-18; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Otologic Disease
Keywords: aprepitant; nausea; vomiting; otologic surgery
MeSH Terms: conditions — Ear Diseases; Nausea; Vomiting | interventions — Aprepitant

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind placebo-controlled trial will be conducted at a single academic institution (Jewish General Hospital) after approval from the Research Ethics Board.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Arm (Experimental): Oral aprepitant 80mg within an hour of induction
  Interventions: Drug: Aprepitant
- Control Arm (Placebo Comparator): Placebo capsule within an hour of induction
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Aprepitant — Participants will be randomly assigned to the intervention or control group in a 1:1 ratio. Oral aprepitant of 80mg will be administered within an hour of induction for an otological surgery.
  Arms: Treatment Arm
Other: Placebo — Participants will be randomly assigned to the intervention or control group in a 1:1 ratio. An oral placebo capsule will be administered within an hour of induction for an otological surgery.
  Arms: Control Arm

SUMMARY:
This project is being carried out to study the use of a medication to reduce nausea and vomiting after ear surgery.

DETAILED DESCRIPTION:
Post-operative nausea and vomiting (PONV) is one of the most common post-surgical complications and is associated with prolonged hospital stays, higher readmission rates, and heightened physical and emotional burden on patients and their families. While the general incidence of PONV is reported to be approximately 20-30% across all specialties, it may affect up to 60-80% of patients undergoing middle ear surgery. Indeed, surgical drilling and irrigation close to inner ear structures may stimulate the vestibular system and activate the chemoreceptor trigger zone and emetic center.

Aprepitant is a novel selective neurokinin-1 (NK1) antagonist which has been extensively studied for the prevention of chemotherapy-induced nausea and vomiting. Randomized controlled trials in gynecologic and open abdominal surgery have shown pre-operative oral aprepitant may provide benefit in reducing nausea and vomiting in the post-operative setting, even beyond commonly employed anti-emetics such as 5HT3 receptor antagonists4. While some authors have reported on its use in thyroid, facial plastics and transsphenoidal surgery, no trial to date has specifically investigated the use of pre-operative aprepitant as an adjunctive medication to reduce post-operative nausea and vomiting in patients undergoing middle ear surgery.

The hypothesis of this research project is that pre-operative aprepitant will provide the added benefit in reducing the incidence of post-operative nausea and vomiting in patients undergoing middle ear surgery when administered in conjunction with a 5-HT3 antagonist and dexamethasone.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing middle ear surgery including tympanoplasty with or without ossicular chain reconstruction, tympanomastoidectomy or stapedectomy
* Patient using a hormonal contraceptive will be included, but warned aprepitant may reduce the efficacy of hormonal contraception thus an alternative or backup contraceptive methods should be used for one month after surgery

Exclusion Criteria:

* Children (<18 years old)
* Patients unable to complete the post-procedure questionnaire (either due to time constraints, neurocognitive impairment, etc.)
* Patients taking concomitant medications that are substrates, inhibitors or inducers of CYP3A4 or CYP2CP that are at risk of having a clinically significant effect
* Patients with a history of hypersensitivity reaction to any of the medications used in the study
* Patients who are pregnant or breastfeeding
* Patients unable to receive general anesthesia (i.e. procedures performed under local anesthesia with or without sedation)
* Patients with severe hepatic insufficiency (Child-Pugh class C)
* Patients on total intravenous anesthesia (TIVA)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of clinically important postoperative nausea and vomiting | 6h to 48h postoperatively
  Using the Postoperative Nausea and Vomiting Intensity Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Only IPD used in the results publication.